CLINICAL TRIAL: NCT03216265
Title: A Proof of Concept (POC) Clinical Study to Investigate the Effects of a Developmental Cosmetic Moisturising Cream on the Barrier Function of Human Skin on the Face and Forearm
Brief Title: A Proof of Concept Clinical Study to Investigate the Effects of an Experimental Cosmetic Moisturiser on the Barrier Function of Human Skin on the Face and Forearm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207451
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-03

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product/ No treatment (Other): Participants randomized to this arm will apply Test product at allocated sites and leave other sites untreated.
  Interventions: Other: Test product (Moisturising cream); Other: No treatment
- Test product/positive control (Other): Participants randomized to this arm will apply Test and positive product at allocated sites.
  Interventions: Other: Test product (Moisturising cream); Other: Positive control (Commercial market place moisturising cream)
- Positive control /no treatment (Other): Participants randomized to this arm will apply Positive product at allocated sites and leave other sites untreated.
  Interventions: Other: Positive control (Commercial market place moisturising cream); Other: No treatment

INTERVENTIONS:
Other: Test product (Moisturising cream) — Participants will be instructed to apply their assigned product to the randomly assigned sites twice daily (in the morning and evening).
  Arms: Test product/ No treatment; Test product/positive control
Other: Positive control (Commercial market place moisturising cream) — Participants will be instructed to apply their assigned product to the randomly assigned sites twice daily (in the morning and evening).
  Arms: Positive control /no treatment; Test product/positive control
Other: No treatment — No treatment.
  Arms: Positive control /no treatment; Test product/ No treatment

SUMMARY:
The objective of this POC clinical study is to investigate the impact of the test product (Developmental Cosmetic Moisturising Cream) on skin barrier function and skin moisturisation on the forearm and face after 4 weeks of twice daily application compared to no treatment in participants with dry sensitive skin.

DETAILED DESCRIPTION:
Areas on the volar forearm and each side of the face, will be selected for measurements of transepidermal water loss (TEWL) and corneometry to be conducted . A physical challenge and a regression period of 5 days is also included to evaluate skin barrier function and moisturisation.

A regression period of 5 days (Days 30, 31, 32, 33 and 34) of no study product use following the 4 week treatment phase is also included to evaluate skin barrier function and moisturisation.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Self-reported dry, sensitive skin on the face and body.
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits.
* Trained examiner visual grading assessment score (including subject self-assessment of tightness) of overall dryness ≥ 3 with a score of at least 1 in the roughness parameter and 4 (for any individual parameter) on each of the forearms and each side of the face at the Screening visit (Visit 1) and Baseline visit (Visit 2).
* In addition, there will be no greater than 0.5 point difference between trained examiner visual grading scores of each volar forearm and each side of the face at the Screening and Baseline visits.
* Fitzpatrick skin type I-IV

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluations.
* Presence of open sores, pimples, or cysts at the application site.
* Active dermatosis (local or disseminated) that might interfere with the results of the study.
* Considered immune compromised.
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the subject at undue risk.
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before screening visit.
* Intention of using any oral or topical steroids.
* Regular use of inhaled steroids (occasional use is permitted).
* Regular use of topical anti-itch medications (occasional use permitted; the product should be applied with an applicator but not to the proposed application areas.
* Use of any topical drug or medication in the proposed application areas.
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit.
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation.
* Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication.
* Known or suspected intolerance or hypersensitivity to any of the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 14 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* Smoker (including e-cigarettes)
* Moles, tattoos, scars, hairs, etc. at the test areas if it is likely that they could affect the assessments.
* Subject has visible sunburn on the test sites.
* Use of self-tanning products on the test areas (face and arms) within 2 weeks prior to the screening visit.
* Any individual parameter score 4 on any test areas of the face or either of the forearms as assessed by a trained examiner.
* Any Subject who, in the judgment of the Investigator, should not participate in the study.
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 69 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nisbet S, Mahalingam H, Gfeller CF, Biggs E, Lucas S, Thompson M, Cargill MR, Moore D, Bielfeldt S. Cosmetic benefit of a biomimetic lamellar cream formulation on barrier function or the appearance of fine lines and wrinkles in randomized proof-of-concept clinical studies. Int J Cosmet Sci. 2019 Feb;41(1):1-11. doi: 10.1111/ics.12499. Epub 2019 Feb 22. PMID 30414275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at one center in Germany.
Pre-assignment Details: A total of 93 participants were screened, out of which 24 did not meet study criteria. Remaining 69 participants were enrolled in the study, out of which 3 did not start the study. 2 were lost to follow-up and 1 due to other reason (not specified).
Groups:
- No Treatment/ Test Product: Participants randomized to this arm applied Test product at allocated side and left other sites untreated.
- No Treatment/ Positive Control: Participants randomized to this arm applied Positive product at allocated sites and left other side untreated.
- Test Product/ Positive Control: Participants randomized to this arm applied Test and positive product at allocated side.
Period: Overall Study
Arm/Group | No Treatment/ Test Product | No Treatment/ Positive Control | Test Product/ Positive Control
Started | 22 | 22 | 22
Completed | 20 | 21 | 19
Not Completed | 2 | 1 | 3
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who applied any of the study products.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment/ Test Product | No Treatment/ Positive Control | Test Product/ Positive Control | Total
Number analyzed (Participants) | 22 | 22 | 22 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 22 | 66
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 22 | 66
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 22 | 22 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) Measurements on Day 29, Test Product Treated Versus (vs.) Untreated Sites on the Forearm
Description: TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 seconds (sec), to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: At Baseline and Day 29
Population: Analysis population was Intent To Treat (ITT) (N=65) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available. Number of participants analyzed for this outcome measure were part of the ITT population, evaluated on Day 29.
Measure: Mean (Standard Deviation); unit: gram (g)/meter(m)^2/hour
Groups:
- Test Product: Data of this arm included all allotted sides of the face of the participants where test product was applied during the study.
- No Treatment: Data of this arm included all allotted sides of the face of the participants which were left untreated during the study.
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 40 | 42
gram (g)/meter(m)^2/hour | -0.59 (2.005) | 0.79 (1.555)
Statistical Analysis 1: Comparison: Test Product vs No Treatment; Test type: Other; p < 0.0001, ANCOVA; Analysis model (ANCOVA) included participant as random effect, treatment arm and side of body as fixed effects, and baseline value as covariate; Least Square Mean difference = -1.44, 95% CI 2-sided [-2.10 to -0.78] — Difference is the first named treatment adjusted (LS) mean change from baseline (Visit 2) minus the second named treatment adjusted mean change from baseline (Visit 2)

2. Secondary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) Measurements on Day 29, Test Product Treated vs. Untreated Sites on the Face
Description: TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: At Baseline and Day 29
Population: Analysis population was ITT (N=65) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available. Number of participants analyzed for this outcome measure were part of the ITT population, evaluated on Day 29.
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 40 | 42
g/m^2/hour | -4.33 (3.729) | -3.18 (3.841)

3. Secondary Outcome: Change From Baseline in Corneometry on the Forearm and Face, Test Product Treated vs. Untreated Sites
Description: Corneometry was used to measure moisture content of stratum corneum using corneometer. The measuring principle is based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. The Corneometer measurements was taken 5 times in total and then an average reading was calculated for each site and time point. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: At Baseline, Day 1 (30 minutes and 6 hours post study product application), Day 2, 15, and 29
Population: Analysis population was ITT (N=65) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available. Here, number analyzed signifies number of participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: Corneometry Units
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
Corneometry Units
  Day 1 (30 mins), change from baseline forearm | 14.29 (6.227) | -3.24 (5.556)
  Day 1 (6 hours), change from baseline, forearm | 10.72 (5.174) | -0.34 (4.908)
  Day 2, change from baseline, forearm | 8.65 (5.954) | 1.48 (4.310)
  Day 15, change from baseline, forearm: number analyzed (Participants) | 41 | 41
  Day 15, change from baseline, forearm | 12.02 (7.149) | 3.06 (5.343)
  Day 29, change from baseline, forearm: number analyzed (Participants) | 40 | 42
  Day 29, change from baseline, forearm | 11.85 (8.665) | 4.50 (6.498)
  Day 1 (30 mins) change from baseline, face | 25.12 (9.093) | -6.96 (7.647)
  Day 1 (6 hours ), change from baseline, face | 13.94 (7.634) | -1.90 (7.152)
  Day 2, change from baseline, face | 8.88 (8.501) | -0.45 (7.867)
  Day 15, change from baseline, face: number analyzed (Participants) | 41 | 41
  Day 15, change from baseline, face | 13.92 (9.976) | 2.50 (12.227)
  Day 29, change from baseline, face: number analyzed (Participants) | 40 | 42
  Day 29, change from baseline, face | 16.94 (10.193) | 3.81 (11.580)

4. Secondary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) on the Forearm and Face, Test Product Treated vs. Untreated Sites at Day 2 and 15
Description: as for outcome 2
Time Frame: At Baseline, Day 2, and 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
g/m^2/hour
  Day 2, change from baseline, forearm | 0.08 (1.766) | 0.48 (1.458)
  Day 15, change from baseline, forearm: number analyzed (Participants) | 41 | 41
  Day 15, change from baseline, forearm | -0.23 (2.874) | 1.07 (2.515)
  Day 2, change from baseline, face | -1.49 (2.624) | 0.77 (3.969)
  Day 15, change from baseline, face: number analyzed (Participants) | 41 | 41
  Day 15, change from baseline, face | -4.79 (3.895) | -2.37 (4.354)

5. Secondary Outcome: Standardised Area Under Curve (AUC1-29) of Change From Baseline in Corneometry Over Treatment Period
Description: Standardised AUC1-29 was calculated for each participant for change from baseline in corneometry on forearms and face over the treatment period; i.e. up to Day 29 using the trapezoidal rule and dividing by the number of days in the period. Corneometry was used to measure moisture content of stratum corneum using corneometer. The measuring principle is based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. The Corneometer measurements was taken 5 times in total and then an average reading was calculated for each site and time point. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: Up to Day 29
Population: Analysis population was ITT (N=65) population included all participants who were randomized into the study and had at least one post-baseline clinical assessment available. Here, number analyzed signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Corneometry units
Groups:
- Positive Control: Data of this arm included all allotted sides of the face of the participants where positive control was applied during the study.
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
Corneometry units
  AUC1-29, Forearm: number analyzed (Participants) | 39 | 40 | 41
  AUC1-29, Forearm | 10.87 (5.732) | 10.20 (6.043) | 2.88 (4.028)
  AUC1-29, Face: number analyzed (Participants) | 39 | 40 | 41
  AUC1-29, Face | 14.03 (7.061) | 15.90 (10.719) | 2.05 (9.149)

6. Secondary Outcome: Standardised Area Under Curve (AUC1-29) of Change From Baseline in Transepidermal Water Loss (TEWL) Over Treatment Period
Description: Standardised AUC1-29 was calculated for each participant for change from baseline in TEWL on forearms and face over the treatment period; i.e. up to Day 29 using the trapezoidal rule and dividing by the number of days in the period. TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Up to Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | Positive Control | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
g/m^2/hour
  AUC1-29, Forearm: number analyzed (Participants) | 39 | 40 | 41
  AUC1-29, Forearm | -0.30 (1.849) | -0.42 (1.572) | 0.82 (1.465)
  AUC1-29, Face: number analyzed (Participants) | 39 | 40 | 41
  AUC1-29, Face | -3.95 (2.950) | -3.21 (4.465) | -1.67 (2.998)

7. Secondary Outcome: Change From Pre-challenge in Transepidermal Water Loss (TEWL) Measurements of D-Squame Discs Following 4, 8 and 12 Adhesive Discs Removal From Skin of Both Test Product Treated and Untreated Sites on the Forearm on Day 29
Description: A series of D-Squame discs were gently smoothed over the designated D-Squame Areas by applying a uniform pressure for 5 secs with a stamp to ensure consistent adhesion to the skin. Each disc was pulled off the skin with one fluent and decisive movement. There were maximum of 12 D-Squame discs (in groups of 4) removed from each forearm repeatedly. TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. TEWL was measured pre-challenge and after 4, 8 and 12 discs have been removed from the forearms. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: On Day 29 (including Pre-challenge)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
g/m^2/hour
  Pre-challenge Day 29: number analyzed (Participants) | 40 | 42
  Pre-challenge Day 29 | 6.96 (1.513) | 8.33 (2.307)
  Change from pre-challenge after 4 discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 4 discs | 2.60 (1.504) | 3.06 (1.995)
  Change from pre-challenge after 8 discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 8 discs | 3.35 (1.662) | 4.94 (3.564)
  Change from pre-challenge after 12 discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 12 discs | 5.56 (2.780) | 8.46 (6.392)

8. Secondary Outcome: Change From Pre-challenge in Transepidermal Water Loss (TEWL) Measurements of D-Squame Discs Following 3, 6 and 9 Adhesive Discs Removal From Skin of Both Test Product Treated and Untreated Sites on the Face on Day 29
Description: A series of D-Squame discs were gently smoothed over the designated D-Squame Areas by applying a uniform pressure for 5 secs with a stamp to ensure consistent adhesion to the skin. Each disc was pulled off the skin with one fluent and decisive movement. There were maximum of 9 D-Squame discs (in groups of 3) removed from the face repeatedly. TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. TEWL was measured pre-challenge and after 3, 6 and 9 discs have been removed from the face. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: On Day 29 (including Pre-challenge)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
g/m^2/hour
  Pre-challenge Day 29: number analyzed (Participants) | 40 | 42
  Pre-challenge Day 29 | 13.10 (4.424) | 14.63 (5.698)
  Change from pre-challenge after 3 Discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 3 Discs | 4.58 (3.261) | 6.45 (4.531)
  Change from pre-challenge after 6 Discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 6 Discs | 11.34 (6.102) | 16.66 (10.636)
  Change from pre-challenge after 9 Discs: number analyzed (Participants) | 40 | 42
  Change from pre-challenge after 9 Discs | 20.68 (12.242) | 27.26 (15.987)

9. Secondary Outcome: Protein Analysis (SquameScan) of D-Squame Discs (Total of 12 Adhesive Discs) From Skin of Both Test Product Treated and Untreated Sites on the Forearm on Day 29
Description: The protein content of each D-Squame disc was analysed using a SquameScan. SquameScan is the instrument used to indirectly measure the protein content extracted from the skin by D-squame tape strips. The determination was performed by measuring the optical absorption of the strip at about 850 nanometres (nm) (infrared light). The value displayed in % was proportionally related to the protein content. The protein content was analysed for each of the discs obtained the D-Squame stripping on the forearms and reported to 2 decimal places.
Time Frame: On Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 40 | 42
Percent | 173.16 (44.816) | 213.89 (29.648)

10. Secondary Outcome: Protein Analysis of D-Squame Discs (Total of 9 Adhesive Discs) From Skin of Both Test Product Treated and Untreated Sites on the Face on Day 29
Description: The protein content of each D-Squame disc was analysed using a SquameScan. SquameScan is the instrument used to indirectly measure the protein content extracted from the skin by D-squame tape strips. The determination was performed by measuring the optical absorption of the strip at about 850 nm (infrared light). The value displayed in % was proportionally related to the protein content. The protein content was analysed for each of the discs obtained the D-Squame stripping on the face and reported to 2 decimal places.
Time Frame: On Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of absorption
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 40 | 42
percent of absorption | 84.70 (23.413) | 107.75 (20.999)

11. Secondary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) Measurements on Days 30, 31, 32, 33 and 34 in Test Product Treated vs. Untreated Sites on the Forearm and Face
Description: TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value was established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: At Baseline, Day 30, 31, 32, 33 and 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 41
g/m^2/hour
  Day 30, Change from baseline, forearm: number analyzed (Participants) | 38 | 40
  Day 30, Change from baseline, forearm | -0.37 (2.351) | 1.12 (2.348)
  Day 31, Change from baseline, forearm: number analyzed (Participants) | 37 | 41
  Day 31, Change from baseline, forearm | -0.77 (1.986) | 1.53 (2.804)
  Day 32,Change from baseline, forearm: number analyzed (Participants) | 39 | 41
  Day 32,Change from baseline, forearm | -0.17 (2.322) | 1.48 (2.110)
  Day 33,Change from baseline, forearm: number analyzed (Participants) | 37 | 40
  Day 33,Change from baseline, forearm | -0.42 (1.902) | 1.00 (1.961)
  Day 34, Change from baseline, forearm: number analyzed (Participants) | 39 | 41
  Day 34, Change from baseline, forearm | -0.59 (1.889) | 1.18 (1.927)
  Day 30, Change from baseline, face: number analyzed (Participants) | 38 | 40
  Day 30, Change from baseline, face | -4.40 (4.145) | -3.18 (3.873)
  Day 31, Change from baseline, face: number analyzed (Participants) | 37 | 41
  Day 31, Change from baseline, face | -4.26 (4.787) | -3.27 (4.112)
  Day 32, Change from baseline, face: number analyzed (Participants) | 39 | 41
  Day 32, Change from baseline, face | -3.27 (5.264) | -3.05 (4.672)
  Day 33, Change from baseline, face: number analyzed (Participants) | 37 | 40
  Day 33, Change from baseline, face | -3.52 (4.781) | -3.64 (3.736)
  Day 34, Change from baseline, face: number analyzed (Participants) | 39 | 41
  Day 34, Change from baseline, face | -3.52 (4.941) | -3.18 (4.035)

12. Secondary Outcome: Change From Day 29 in Transepidermal Water Loss (TEWL) Measurements on Days 30, 31, 32, 33 and 34 in Test Product Treated vs. Untreated Sites on the Forearm and Face
Description: as for outcome 11
Time Frame: At Day 30, 31, 32, 33, and 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
g/m^2/hour
  Day 30, change from Day 29, forearm: number analyzed (Participants) | 38 | 40
  Day 30, change from Day 29, forearm | 0.20 (1.970) | 0.25 (1.696)
  Day 31, change from Day 29, forearm: number analyzed (Participants) | 37 | 41
  Day 31, change from Day 29, forearm | -0.09 (1.494) | 0.72 (1.885)
  Day 32, change from Day 29, forearm: number analyzed (Participants) | 39 | 41
  Day 32, change from Day 29, forearm | 0.45 (1.962) | 0.67 (1.444)
  Day 33, change from Day 29, forearm: number analyzed (Participants) | 37 | 40
  Day 33, change from Day 29, forearm | 0.26 (1.673) | 0.19 (1.737)
  Day 34, change from Day 29, forearm: number analyzed (Participants) | 39 | 41
  Day 34, change from Day 29, forearm | 0.03 (1.669) | 0.37 (1.649)
  Day 30, change from Day 29, face: number analyzed (Participants) | 38 | 40
  Day 30, change from Day 29, face | 0.10 (3.341) | -0.05 (2.000)
  Day 31, change from Day 29, face: number analyzed (Participants) | 37 | 41
  Day 31, change from Day 29, face | 0.22 (3.807) | 0.01 (2.833)
  Day 32, change from Day 29, face: number analyzed (Participants) | 39 | 41
  Day 32, change from Day 29, face | 1.17 (4.399) | 0.22 (2.941)
  Day 33, change from Day 29, face: number analyzed (Participants) | 37 | 40
  Day 33, change from Day 29, face | 1.00 (3.454) | -0.41 (2.286)
  Day 34, change from Day 29, face: number analyzed (Participants) | 39 | 41
  Day 34, change from Day 29, face | 0.91 (4.047) | 0.09 (2.594)

13. Secondary Outcome: Change From Baseline in Standardised Area Under Curve (AUCday 29-34) of Transepidermal Water Loss (TEWL) Over Regression Period (Days 30, 31, 32, 33 and 34) of Forearm and Face, Test Product Treated vs. Untreated Sites
Description: Standardised AUCday29-34 was calculated for each participant for change from baseline in TEWL on forearms and face over the regression period (Day31, 32, 33 and 34) using the trapezoidal rule and dividing by the number of days in the period. TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value was established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Up to Day 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Groups:
- Test Product: Data of this arm included all allotted sides of the face of the participant where test product was applied during the study.
- No Treatment: Data of this arm included all allotted sides of the face of the participant which were left untreated during the study.
Arm/Group | Positive Control | Test Product | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
g/m^2/hour
  Change from baseline in AUCday29-34, forearm: number analyzed (Participants) | 38 | 35 | 39
  Change from baseline in AUCday29-34, forearm | -0.51 (3.033) | -0.54 (1.777) | 1.25 (1.897)
  Change from baseline in AUCday29-34, face: number analyzed (Participants) | 43 | 35 | 39
  Change from baseline in AUCday29-34, face | -4.81 (4.329) | -3.94 (4.187) | -3.21 (3.917)

14. Secondary Outcome: Change From Day 29 in Standardised Area Under Curve (AUCday 29-34) of Transepidermal Water Loss (TEWL) Over Regression Period (Days 30, 31, 32, 33 and 34) of Forearm and Face, Test Product Treated vs. Untreated Sites
Description: Standardised AUCday29-34 was calculated for each participant for change from Day 29 in TEWL on forearms and face over the regression period (Day31, 32, 33 and 34) using the trapezoidal rule and dividing by the number of days in the period. TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value was established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 secs were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Up to Day 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Positive Control | Test Product | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
g/m^2/hour
  Change from Day 29 in AUCday29-34, forearm: number analyzed (Participants) | 38 | 35 | 39
  Change from Day 29 in AUCday29-34, forearm | 0.66 (2.166) | 0.13 (1.296) | 0.38 (1.056)
  Change from Day 29 in AUCday29-34, face: number analyzed (Participants) | 38 | 35 | 39
  Change from Day 29 in AUCday29-34, face | 0.38 (2.114) | 0.51 (3.006) | -0.13 (1.980)

15. Secondary Outcome: Change From Baseline in Corneometry Measurements on Days 30, 31, 32, 33 and 34 in Test Product Treated Site vs. Untreated Site on the Forearm and Face
Description: Corneometry was used to measure the moisture content of stratum corneum using corneometer. The measuring principle is based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. The Corneometer measurements were taken 5 times in total and then an average reading was calculated for each site and time point. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: At Baseline, Day 30, 31, 32, 33, and 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Corneometry units
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
Corneometry units
  Day 30, change from baseline, forearm: number analyzed (Participants) | 38 | 40
  Day 30, change from baseline, forearm | 7.11 (7.862) | 3.48 (6.298)
  Day 31,change from baseline, forearm: number analyzed (Participants) | 37 | 41
  Day 31,change from baseline, forearm | 5.51 (7.653) | 3.54 (6.652)
  Day 32,change from baseline, forearm: number analyzed (Participants) | 39 | 41
  Day 32,change from baseline, forearm | 4.25 (8.419) | 2.25 (6.639)
  Day 33,change from baseline, forearm: number analyzed (Participants) | 37 | 40
  Day 33,change from baseline, forearm | 2.85 (7.444) | 1.54 (6.645)
  Day 34,change from baseline, forearm: number analyzed (Participants) | 39 | 41
  Day 34,change from baseline, forearm | 3.53 (10.071) | 1.99 (8.216)
  Day 30,change from baseline, face: number analyzed (Participants) | 38 | 40
  Day 30,change from baseline, face | 9.68 (8.772) | 2.35 (11.473)
  Day 31,change from baseline, face: number analyzed (Participants) | 37 | 41
  Day 31,change from baseline, face | 7.40 (8.909) | 0.76 (10.885)
  Day 32,change from baseline, face: number analyzed (Participants) | 39 | 41
  Day 32,change from baseline, face | 5.93 (8.382) | 0.41 (10.749)
  Day 33,change from baseline, face: number analyzed (Participants) | 37 | 40
  Day 33,change from baseline, face | 2.93 (7.597) | -2.38 (10.834)
  Day 34,change from baseline, face: number analyzed (Participants) | 39 | 41
  Day 34,change from baseline, face | 4.76 (11.119) | 1.09 (12.370)

16. Secondary Outcome: Change From Day 29 in Corneometry Measurements on Days 30, 31, 32, 33 and 34 in Test Product Treated Site vs. Untreated Site on the Forearm and Face
Description: as for outcome 15
Time Frame: At Day 29, 30, 31, 32, 33, and 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Corneometry units
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 43 | 44
Corneometry units
  Day 30, change from Day 29, forearm: number analyzed (Participants) | 38 | 40
  Day 30, change from Day 29, forearm | -4.44 (4.913) | -1.06 (5.376)
  Day 31,change from Day 29, forearm: number analyzed (Participants) | 37 | 41
  Day 31,change from Day 29, forearm | -6.37 (4.788) | -1.10 (3.724)
  Day 32,change from Day 29, forearm: number analyzed (Participants) | 39 | 41
  Day 32,change from Day 29, forearm | -7.72 (4.903) | -2.38 (5.634)
  Day 33,change from Day 29, forearm: number analyzed (Participants) | 37 | 40
  Day 33,change from Day 29, forearm | -8.63 (4.716) | -3.02 (5.590)
  Day 34,change from Day 29, forearm: number analyzed (Participants) | 39 | 41
  Day 34,change from Day 29, forearm | -8.43 (6.539) | -2.65 (6.933)
  Day 30,change from Day 29, face: number analyzed (Participants) | 38 | 40
  Day 30,change from Day 29, face | -7.84 (7.647) | -1.57 (7.307)
  Day 31,change from Day 29, face: number analyzed (Participants) | 37 | 41
  Day 31,change from Day 29, face | -9.59 (7.999) | -3.09 (6.784)
  Day 32,change from Day 29, face: number analyzed (Participants) | 39 | 41
  Day 32,change from Day 29, face | -11.28 (8.316) | -3.44 (7.539)
  Day 33,change from Day 29, face: number analyzed (Participants) | 37 | 40
  Day 33,change from Day 29, face | -14.22 (8.466) | -6.15 (8.095)
  Day 34,change from Day 29, face: number analyzed (Participants) | 39 | 41
  Day 34,change from Day 29, face | -12.45 (11.925) | -2.77 (8.020)

17. Secondary Outcome: Standardised Area Under Curve (AUCday29-34) Calculated Using Change From Baseline in Corneometry Over Regression Period (Days 30, 31, 32, 33 and 34) on the Forearm and Face
Description: Standardised AUCday29-34 was calculated for each participant for change from baseline in corneometry on forearms and face over the regression period using the trapezoidal rule and dividing by the number of days in the period. Corneometry was used to measure moisture content of stratum corneum using corneometer. The measuring principle is based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. The Corneometer measurements was taken 5 times in total and then an average reading was calculated for each site and time point. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: Up to Day 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Corneometry units
Arm/Group | Positive Control | Test Product | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
Corneometry units
  Change from baseline in AUCday29-34, forearm: number analyzed (Participants) | 43 | 35 | 39
  Change from baseline in AUCday29-34, forearm | 4.12 (6.675) | 4.87 (7.211) | 2.65 (5.999)
  Change from baseline in AUCday29-34, face: number analyzed (Participants) | 38 | 35 | 39
  Change from baseline in AUCday29-34, face | 7.01 (10.824) | 7.21 (7.427) | 0.84 (10.386)

18. Secondary Outcome: Standardised AUC Calculated Using Change From Day 29 in Corneometry Over Regression Period (Days 30, 31, 32, 33 and 34) on the Forearm and Face
Description: Standardised AUCday29-34 was calculated for each participant for change from day 29 in corneometry on forearms and face over the regression period using the trapezoidal rule and dividing by the number of days in the period. Corneometry was used to measure the moisture content of stratum corneum using corneometer. The measuring principle is based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. The Corneometer measurements were taken 5 times in total and then an average reading was calculated for each site and time point. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: Up to Day 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Corneometry units
Arm/Group | Positive Control | Test Product | No Treatment
Number analyzed (Participants) | 43 | 43 | 44
Corneometry units
  Change from Day 29 in AUCday29-34, forearm: number analyzed (Participants) | 38 | 35 | 39
  Change from Day 29 in AUCday29-34, forearm | -5.34 (3.197) | -6.24 (3.642) | -1.81 (4.065)
  Change from Day 29 in AUCday29-34, face: number analyzed (Participants) | 38 | 35 | 39
  Change from Day 29 in AUCday29-34, face | -11.56 (6.726) | -10.04 (6.804) | -2.99 (5.586)

19. Secondary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) Measurements on Day 29 of Positive Control Treated Site vs. Untreated Site on the Forearm.
Description: TEWL measuring principle is based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 secs, to ensure that a stable value has been established. The first part of the measurement belongs to the equilibration phase. The values of the last 10 seconds were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: At Baseline and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/m^2/hour
Arm/Group | Positive Control | No Treatment
Number analyzed (Participants) | 40 | 42
g/m^2/hour | -1.13 (2.104) | 0.79 (1.555)

ADVERSE EVENTS:
Time Frame: Approximately 42 days.
Description: All treatment emergent adverse events (AEs) were reported in this section. Skin-related AEs counted under one or both treatment groups that the participants received based on the application site(s). Non-skin related adverse events counted under both treatment groups that the participant received. Each adverse event was counted only once in the Overall column irrespective of whether it was skin related or not.
Groups:
- Overall Participants: Included all participants who applied any of the study products.
Arm/Group | Test Product | Positive Control | No Treatment | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/66
Other Adverse Events (participants affected / at risk) | 10/44 | 11/44 | 12/44 | 20/66
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=44) | Positive Control (N=44) | No Treatment (N=44) | Overall Participants (N=66)
PYREXIA (General disorders) | 2 | 1 | 1 | 2
APPLICATION SITE ERYTHEMA (General disorders) | 1 | 0 | 2 | 2
APPLICATION SITE PAPULES (General disorders) | 1 | 2 | 0 | 3
APPLICATION SITE PRURITUS (General disorders) | 1 | 0 | 1 | 2
APPLICATION SITE SCAB (General disorders) | 1 | 0 | 1 | 1
APPLICATION SITE BURN (General disorders) | 0 | 1 | 0 | 1
APPLICATION SITE DRYNESS (General disorders) | 0 | 1 | 0 | 1
APPLICATION SITE PAIN (General disorders) | 0 | 1 | 0 | 1
APPLICATION SITE REACTION (General disorders) | 0 | 0 | 1 | 1
INJURY ASSOCIATED WITH DEVICE (General disorders) | 0 | 0 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 1 | 3 | 4
CYSTITIS (Infections and infestations) | 1 | 1 | 0 | 1
EAR INFECTION (Infections and infestations) | 1 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 4 | 3 | 5
MIGRAINE (Nervous system disorders) | 1 | 2 | 1 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 1 | 1
NEPHRITIS (Renal and urinary disorders) | 1 | 1 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
EYELID OEDEMA (Eye disorders) | 1 | 0 | 1 | 1
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 1 | 1
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT03216265/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03216265/SAP_001.pdf